CLINICAL TRIAL: NCT03821831
Title: Residual Pediatric Obstructive Sleep Apnea: Closing the Treatment Gap
Brief Title: Treating Children With Obstructive Sleep Apnea After Surgery Failure
Status: Terminated | Type: Observational
Why Stopped: COVID hindered enrollment
Sponsor: University of Alberta (Other)
Collaborators: Natural Sciences and Engineering Research Council, Canada (Other)
Responsible Party: Sponsor
Other Study IDs: GHeo
Record Dates: First submitted 2019-01-10; First posted 2019-01-30 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Pediatric Obstructive Sleep Apnea; Pediatric Obesity
Keywords: Obstructive sleep apnea; Children; Orthodontic intervention; Nutrition; Metabolomic markers
MeSH Terms: conditions — Pediatric Obesity; Sleep Apnea, Obstructive | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine, blood and saliva
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (3):
- Continuous Positive Airway Pressure: This group consists of consenting patients and their parents who choose Continuous Positive Airway Pressure (CPAP). The CPAP is a type of therapy that applies mild air pressure to a person's upper airway to keep their airway open so that they can breathe normally while they sleep.
  Interventions: Device: Continuous Positive Airway Pressure
- Orthodontic Intervention: This group consists of consenting patients and their parents who choose orthodontic intervention will be seen by participating orthodontists who will determine types of orthodontic intervention; mandibular advancement devices or rapid maxillary expansion devices, or Class III mid face advancement with skeletal anchored headgear. In this group, the patients will also receive a biometric shirt to use once every two weeks, to monitor their sleep during the study.
  Interventions: Device: Orthodontic intervention
- Control: This group consists of consenting patients and their parents who choose to remain untreated. In this group, the patients will also receive a biometric shirt to use once every two weeks, to monitor their sleep during the study.

INTERVENTIONS:
Device: Continuous Positive Airway Pressure — CPAP machine
  Groups: Continuous Positive Airway Pressure
Device: Orthodontic intervention — Mandibular advancement or Rapid maxillary expansion devices
  Groups: Orthodontic Intervention

SUMMARY:
The aim of this study is to evaluate the potential improvement of sleep quality in children who have residual obstructive sleep apnea, using either an orthodontic intervention or continuous positive airway pressure (CPAP), versus no treatment.

DETAILED DESCRIPTION:
Consenting patients and their parents will choose one of three options (within the context of medical/craniofacial appropriateness): CPAP, orthodontic intervention, or to remain untreated (control). It would be ideal if each patient was randomly assigned to one of three groups. However, in our study, random allocation is not an option as the established clinical pathways for treatment, financial resources, and physiological presentation of the patient determines the appropriate intervention. In each group, the effectiveness of the intervention will be analyzed through the evaluation of sleep parameters, medical history, questionnaire responses, craniofacial characteristics, diet, and metabolomic markers, each at baseline and at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with obstructive sleep apnea by polysomnography who presented with a failure in treatment with surgical removal of the tonsils and adenoid tissue --adenotonsillectomy (T&A).
* Patients diagnosed with obstructive sleep apnea but for whom T&A was not an option following assessment by Otolaryngology.

Exclusion Criteria:

* Autism spectrum
* Down syndrome
* Pulmonary hypertension
* Cystic fibrosis

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children from 6 to16 years old, from both sexes in Alberta, Canada, diagnosed with (a) residual OSA (post-T&A) or (b) diagnosed with OSA but for whom T&A is not a treatment option.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2021-12-03 (Actual); Primary Completion 2023-05-08 (Actual); Study Completion 2023-05-08 (Actual)

PRIMARY OUTCOMES:
Measure of change in OSA severity | baseline and 12 months
  Change from baseline Apnea-Hypopnea Index (OSA severity index) measurement by polysomnography at 12 months
Change from baseline total score Pediatric Sleep Questionnaire (PSQ) at 12 months | baseline and 12 months
  PSQ consists of total 22 questions with choices of answer; Yes or No. Yes answer will be coded as 1 and No answer coded as 0. Sum of 22 questions will be compared.

SECONDARY OUTCOMES:
Change from baseline body mass index (BMI) at 12 months | baseline and 12 months
  Height (m) and weight (kg) will be measured to calculate BMI (kg/m^2).

CONTACTS AND LOCATIONS:
Overall Officials: Giseon Heo, Principal Investigator — Dentistry, University of Alberta; Rochelle Young, Study Chair — Pediatric Respiratory Medicine, University of Alberta Hospital; Paul Major, Study Director — Dentistry, University of Alberta
Locations (1):
- Faculty of Medicine and Dentistry, Edmonton, Alberta, Canada

REFERENCES:
- [Derived] Fagundes NCF, Perez-Garcia A, Graf D, Flores-Mir C, Heo G. Orthodontic interventions as a management option for children with residual obstructive sleep apnea: a cohort study protocol. BMJ Open. 2022 Jun 15;12(6):e061651. doi: 10.1136/bmjopen-2022-061651. PMID 35705345